CLINICAL TRIAL: NCT06989437
Title: A Phase 2b/3, Randomized, Double-Blind Study to Investigate the Efficacy, Safety, and Tolerability of Ponsegromab (PF-06946860) Compared With Placebo Both With Background First-Line Chemotherapy in Adult Participants With Cachexia and Metastatic Pancreatic Ductal Adenocarcinoma
Brief Title: A Study to Learn About the Medicine Ponsegromab in Adults With Cancer of the Pancreas Which Has Spread and Caused Significant Body Weight Loss and Fatigue
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C3651021; 2025-522093-36-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2025-05-07; First posted 2025-05-25 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Cachexia; Metastatic Pancreatic Ductal Adenocarcinoma
Keywords: pancreatic cancer; metastatic cancer; cancer; anorexia; cachexia; weight loss; loss of appetite; fatigue
MeSH Terms: conditions — Cachexia; Pancreatic Neoplasms; Neoplasm Metastasis; Neoplasms; Anorexia; Weight Loss; Fatigue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Double-Blind ponsegromab Treatment lower dose (Experimental): ponsegromab 200 mg subcutaneous injection every 4 weeks
  Interventions: Drug: ponsegromab
- Double-Blind ponsegromab Treatment higher dose (Experimental): ponsegromab 400 mg subcutaneous injection every 4 weeks
  Interventions: Drug: ponsegromab
- Double-Blind Placebo Treatment (Placebo Comparator): Match placebo subcutaneous injection every 4 weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: ponsegromab — Double-Blind ponsegromab Treatment
  Arms: Double-Blind ponsegromab Treatment higher dose; Double-Blind ponsegromab Treatment lower dose
Drug: placebo — Double-Blind placebo Treatment
  Arms: Double-Blind Placebo Treatment

SUMMARY:
Study to investigate the efficacy, safety and tolerability of systemic chemotherapy plus ponsegromab versus systemic chemotherapy plus placebo for the first-line treatment in adult participants with cachexia and metastatic pancreatic ductal adenocardinoma.

DETAILED DESCRIPTION:
A Phase 2b/3, randomized, double-blind, multicenter, multinational study to investigate the efficacy, safety and tolerability of systemic chemotherapy plus ponsegromab versus systemic chemotherapy plus placebo for the first-line treatment in adult participants with cachexia and mPDAC. The first-line chemotherapies will either be nab-paclitaxel plus gemcitabine or FOLFIRINOX (or mFOLFIRINOX). The double-blind period is followed by an optional open-label extension period.

Initial enrollment will be in Phase 2b. If all eligibility criteria are met, participants will be randomized in a 1:1:1 allocation to study intervention (one of the two doses of ponsegromab, or placebo) plus first-line systemic chemotherapy. Participants must have completed their first-line pre-randomization systemic chemotherapy (1 x 28-day cycle of nab-paclitaxel and gemcitabine or 2 x 14-days cycles of FOLFIRINOX) prior to the start of receiving their first dose (Day 1) of study intervention (ponsegromab or placebo). Day 1 study intervention must be taken on the same day participants start their next cycle of nab-paclitaxel and gemcitabine chemotherapy or FOLFIRINOX chemotherapy and prior to receiving chemotherapy. All chemotherapy dosing is to be determined by the participant's health care provider in accordance with local guidelines. Study intervention will be administered Q4W SC.

Following enrollment completion of Phase 2b, Phase 3 enrollment will begin, and eligible participants will be randomized in a 1:1:1 allocation to study intervention (one of the two doses of ponsegromab, or placebo). Participants must have completed their first-line pre-randomization systemic chemotherapy (1 x 28-day cycle of nab-paclitaxel and gemcitabine or 2 x 14-day cycles of FOLFIRINOX) prior to the start of receiving their first dose (Day 1) of study intervention (ponsegromab or placebo). Day 1 study intervention must be taken on the same day participants start their next cycle of nab-paclitaxel and gemcitabine chemotherapy or FOLFIRINOX chemotherapy and prior to receiving chemotherapy. All chemotherapy dosing is to be determined by the participant's health care provider in accordance with local guidelines. Study intervention will be administered Q4W SC.

Once all Phase 2b participants have completed Week 12 procedures, an analysis of Phase 2b will be performed, from which one of the 2 ponsegromab doses will be selected. After the Phase 3 ponsegromab dose has been selected, continuing Phase 2b participants will:

* Continue the ponsegromab dose selected for Phase 3 if already randomized to that dose, OR
* Be switched to the ponsegromab dose selected for Phase 3 if randomized to the non-selected ponsegromab dose, OR
* Continue receiving placebo if randomized to placebo
* Remain blinded to study treatment

After the ponsegromab dose has been selected, continuing Phase 3 participants will:

* Continue the ponsegromab dose selected for Phase 3 if already randomized to that dose, OR
* Be switched to the ponsegromab dose selected for Phase 3 if randomized to the non-selected ponsegromab dose, OR
* Continue receiving placebo if randomized to placebo
* Remain blinded to study treatment Phase 3 participants enrolled after dose selection will be randomized 1:1 (ponsegromab selected dose: placebo). Participants must have completed their first-line pre-randomization systemic chemotherapy (1 x 28-day cycle of nab-paclitaxel and gemcitabine or 2 x 14-days cycles of FOLFIRINOX) prior to the start of receiving their first dose (Day 1) of study intervention (selected Phase 3 ponsegromab dose or placebo). Day 1 study intervention must be taken on the same day participants start their next cycle of nab-paclitaxel and gemcitabine chemotherapy or FOLFIRINOX chemotherapy and prior to receiving chemotherapy.

During the Phase 3 portion of the study, there will be an optional sub-study for primary caregivers of participants with cachexia and mPDAC to evaluate the effectiveness of ponsegromab in improving the quality of life and well-being of the primary caregivers.

Study intervention (ponsegromab selected dose or placebo) will continue regardless of chemotherapy treatment until permanent discontinuation of study intervention, withdrawal of consent, death, or the end of the Phase 3 double-blind portion of the study has been reached when the approximate number of overall survival events have been accrued for the Phase 3 analysis of overall survival.

Participants will have tumor assessments performed approximately every 6 to 8 weeks during the double-blind period by blinded, independent, central reader radiologists.

When the number of overall survival events has been accrued to terminate the Phase 3 double-blind portion of the study, active participants can continue in the optional open-label extension where they will receive ponsegromab for up to 12 months.

ELIGIBILITY:
Key inclusion Criteria:

* Signed Informed Consent Document
* Documented active diagnosis of metastatic pancreatic ductal adenocarcinoma
* Cachexia defined by Fearon criteria of weight loss
* Completed 1 x 28-day cycle of first-line systemic nab-paclitaxel and gemcitabine chemotherapy or 2 x 14-day cycles of FOLFIRINOX chemotherapy and prior to receiving Cycle 2 chemotherapy
* ECOG PS ≤1 with life expectancy of at least 4 months

Key Exclusion Criteria:

* Current active reversible causes of decreased food intake
* Cachexia caused by other reasons
* Any prior or current clinical diagnosis of heart failure, irrespective of left ventricular ejection fraction or New York Heart Association classification
* Left ventricular ejection fraction <50%
* Receiving tube feedings or parenteral nutrition at the time of Screening or Randomization
* History of allergic or anaphylactic reaction to any therapeutic or diagnostic monoclonal antibody
* History of allergy or hypersensitivity to any of the chemotherapeutics or any of their excipients
* Neuroendocrine (carcinoid, islet cell) or acinar pancreatic carcinoma, symptomatic brain metastasis, leptomeningeal disease or other active CNS metastases
* Inadequate liver function
* Renal disease requiring dialysis or eGFR <30 mL/min/1.73m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 982 (Estimated)
Dates: Start 2025-10-03 (Actual); Primary Completion 2028-01-17 (Estimated); Study Completion 2029-12-10 (Estimated)

PRIMARY OUTCOMES:
Percent change from baseline in body weight for ponsegromab compared to placebo | Baseline, Week 12
Change from baseline in Functional Assessment of Anorexia/Cachexia Therapy 5-item Anorexia Symptom Scale scores | Baseline, Week 12
  Scale consists of five items, each rated 0-4. Total score ranges from 0 (minimum) to 20 (maximum). Higher scores are associated with a better outcome.

SECONDARY OUTCOMES:
Change from baseline in non-sedentary physical activity time | Baseline, Week 12
  measured by wearable Digital Health Technology watch
Overall survival | Randomization through completion of Phase 3 of the study, an average of 1 year
  Outcome defined as the time from randomization to occurrence of all-cause death
Change from baseline in body weight (kg) | Baseline, Week 12 and up to Week 52
Change from baseline at Week 12 in physical activity as measured by total vector magnitude | Baseline, Week 12
  measured by wearable Digital Health Technology watch
Effect on progression free survival | Randomization through completion of Phase 3 of the study, an average of 1 year
  determined by Blinded Independent Central Review
Effect on objective response rate | Baseline, Week 52
  determined by Blinded Independent Central Review
Effect on disease control rate | Baseline, Week 52
  determined by Blinded Independent Central Review
Effect on duration of response | Baseline, Week 52
  determined by Blinded Independent Central Review
Change from baseline in skeletal muscle area and radiodensity at third lumbar vertebra (L3) | Baseline, Week 12
  measured by CT (or MRI) scan
Change from baseline in intermuscular adipose area and radiodensity at L3 | Baseline, Week 12
  measured by CT (or MRI) scan
Change from baseline in subcutaneous adipose area and radiodensity at L3 | Baseline, Week 12
  measured by CT (or MRI) scan
Change from baseline in visceral adipose area and radiodensity at L3 | Baseline, Week 12
  measured by CT (or MRI) scan
Number of participants with incidence of Treatment Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), and Adverse Events (AEs) leading to permanent discontinuation from study intervention or from study. | Baseline, Week 12 and up to Week 52
Number of participants with laboratory test abnormalities. | Baseline, Week 12 and up to Week 52
Number of participants with vital signs abnormalities. | Baseline, Week 12 and up to Week 52
Change in physical function, assessed on participant completed Patient-Reported Outcomes Measurement Information System Physical Function (version 8c) questionnaire. | Baseline, Week 12 and up to Week 52
  The overall score range for the T-score is 0-100. Higher scores indicate better outcome.
Change in fatigue, as assessed on participant completed Patient-Reported Outcomes Measurement Information System - Fatigue (version 7a) questionnaire. | Baseline, Week 12 and up to Week 52
  The overall score range for the T-score is 29.4-83.2. Lower scores indicate better outcome.
Occurrence and severity of symptomatic AEs including diarrhea, nausea, vomiting, decreased appetite, fatigue and mouth sores by maximum grade as assessed by the NCI PRO CTCAE. | Baseline, Week 52
Change from baseline on ECOG PS | Baseline, Week 12 and up to Week 52
Occurrence of chemotherapy dosing changes (including dosing reductions, dosing interruptions, and dosing discontinuations) due to occurrence of the TEAEs of nausea, vomiting, diarrhea, loss of appetite, or fatigue | Baseline, up to Week 52
Tumor status | Baseline, Week 12 and up to Week 52
  Assessment of tumor response to treatment as determined by Blinded Independent Central Review assessment per RECIST 1.1 using CT scan (or MRI)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (68):
- United States (19):
  - Central Arkansas Radiation Therapy Institute, dba CARTI, Bryant, Arkansas
  - Central Arkansas Radiation Therapy Institute, dba CARTI, Conway, Arkansas
  - CARTI Cancer Center, Little Rock, Arkansas
  - Central Arkansas Radiation Therapy Institute, dba CARTI, North Little Rock, Arkansas
  - Central Arkansas Radiation Therapy Institute, dba CARTI, Pine Bluff, Arkansas
  - Cedars-Sinai Cancer at Cedars-Sinai Medical Center, Los Angeles, California
  - Providence Medical Foundation, Santa Rosa, California
  - Invision, LLC, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Cardiology Associates, Inc, ‘Aiea, Hawaii
  - Hope and Healing Cancer Services, Hinsdale, Illinois
  - Hope and Healing Cancer Services New Lenox, New Lenox, Illinois
  - Renown Health Medical Oncology, Reno, Nevada
  - Renown Office of Clinical Research, Reno, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - OHSU Center for Health & Healing 1, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - OSHU Center for Health and Healing 2, Portland, Oregon
  - Virginia Mason Medical Center, Seattle, Washington
- Australia (4):
  - Shoalhaven District Memorial Hospital, Nowra, New South Wales
  - ICON Cancer Centre - Kurralta Park, Kurralta Park, South Australia
  - Icon Cancer Centre Hobart, Hobart, Tasmania
  - Western Health-Sunshine & Footscray Hospitals, St Albans, Victoria
- Canada (2):
  - CIUSSS- saguenay-Lac-Saint-Jean, Chicoutimi, Quebec
  - Jewish General Hospital, Montreal, Quebec
- China (2):
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
- India (2):
  - Venkateshwar Hospital, New Delhi, National Capital Territory of Delhi
  - Rajiv Gandhi Cancer Institute And Research Centre, New Delhi, National Capital Territory of Delhi
- Israel (6):
  - Rabin Medical Center, Petah Tikva, Central District
  - Sheba Medical Center, Ramat Gan, Central District
  - Shaare Zedek Medical Center, Jerusalem, Jerusalem
  - Hadassah Medical Center, Jerusalem, Jerusalem
  - Rambam Health Care Campus, Haifa, Northern District
  - Sourasky Medical Center, Tel Aviv, TELL ABĪB
- Japan (14):
  - Chiba cancer center, Chiba, Chiba
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Kagawa University Hospital, Kita-gun, Kagawa-ken
  - St. Marianna University Hospital, Kawasaki, Kanagawa
  - Kanagawa cancer center, Yokohama, Kanagawa
  - The University of Osaka Hospital, Suita, Osaka
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - The Cancer Institute Hospital of JFCR, Koto-ku, Tokyo
  - Wakayama Minami Radiology Clinic, Wakayama-shi Kimiidera 870-2, Wakayama
  - Yamaguchi University Hospital, Ube, Yamaguchi
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Kyushu University Hospital, Fukuoka
  - University Hospital,Kyoto Prefectural University of Medicine, Kyoto
  - Wakayama Medical University Hospital, Wakayama
- Puerto Rico (4):
  - Pan American Center for Oncology Trials, LLC - Dorado Office, Dorado
  - Pan American Center for Oncology Trials, LLC - Mayaguez Office, Mayagüez
  - Pan American Center for Oncology Trials, LLC, Rio Piedras
  - Pan American Center for Oncology Trials, LLC, San Juan
- South Korea (10):
  - Inha University Hospital, Incheon, Incheon-gwangyeoksi [incheon]
  - Seoul National University Bundang Hospital, Seongnam, Kyǒnggi-do
  - CHA Bundang Medical Center, CHA University, Seongnam-si, Kyǒnggi-do
  - Seoul National University Hospital, Seoul, Seoul-teukbyeolsi [seoul]
  - Severance Hospital, Yonsei University Health System, Seoul, Seoul-teukbyeolsi [seoul]
  - Asan Medical Center, Seoul, Seoul-teukbyeolsi [seoul]
  - Samsung Medical Center, Seoul, Seoul-teukbyeolsi [seoul]
  - The Catholic Univ. of Korea Seoul St. Mary's Hospital, Seoul, Seoul-teukbyeolsi [seoul]
  - Keimyung University Dongsan Hospital, Daegu, Taegu-kwangyǒkshi
  - Inje University Haeundae Paik Hospital, Busan
- Taiwan (5):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3651021